CLINICAL TRIAL: NCT04269681
Title: Renovate Palliative Study: Randomized Controlled Trial Comparing High Flow Nasal Catheter Versus Standard Respiratory Support in Patients With Do Not Intubate Order and Acute Respiratory Failure
Brief Title: RENOVATE Palliative: HFNC vs. Standard Respiratory Support in Patients With Do-Not-Intubate Order and ARF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impacted by the COVID-19 pandemic:
  * slow recruitment rate
  * cuts in budget for non-COVID-19 related projects
Sponsor: Hospital do Coracao (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP-HCOR/RENOVATEpaliativo
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Care, Palliative; Respiratory Failure
Keywords: non invasive ventilation; high flow nasal cannula; palliative; dypnea; standard care; do-not-intubate; acute respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Participants will be randomised for 2 groups: high flow nasal cannula or standard care with no crossover between them.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will have no access to randomisation list and won't be able to guess which group participant was allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula Arm (Experimental): Participants will receive HFNC if they have no delirium and signs of ARF. The device is supposed to be used continuously in the nose with some changes in flow and/or temperature according to tolerance. There is no crossover to the standar of care arm.
  Interventions: Device: High Flow Nasal Cannula
- Standard respiratory support (Active Comparator): Participants will receive standard of care with low flow oxygen catheter or mask initially. If there is any sign of clinical deterioration NIV can be offered if tolerated by the patient. There will be no cross over with HFNC arm.
  Interventions: Other: Standard respiratory support

INTERVENTIONS:
Device: High Flow Nasal Cannula — Experimental intervention (HFNC) The HFNC (AIRVO 2 - Fisher & Paykel Healthcare, Auckland, New Zealand) consists of a device that allows FiO2 adjustable from 21 to 100% and that delivers a flow of humidified and heated gas up to 60 l / min and 37 degrees C of temperature.
  The HFNC will be offered until resolution of the ARF or until decision by the assisting team and the patient and/or their legal guardian, for the suspension of the treatment due to intolerance, and/or worsening of the discomfort and / or dyspnea.
  The HFNC should be offered to the patient in ARF as follows:
  * Initial parameters: Flow 45 ml / L, FiO2 50%, AIRVO 37oC temperature;
  * Titrate the flow up to 60ml / L or up to the maximum tolerated;
  * Titrate FiO2 to maintain SatO2 between 92% to 98%, starting with 50%;
  * Keep the AIRVO temperature at 37oC, if not possible, acceptable down to 34oC.
  Other Names: High Flow Oxygen; Airvo; Optiflow; Nasal High Flow
  Arms: High Flow Nasal Cannula Arm
Other: Standard respiratory support — The patient randomized to standard respiratory support will be placed on conventional low flow oxygen therapy according to the center's standard of care aiming at SpO2 90 - 98% and improvement of dyspnea. For cases refractory to oxygen therapy, keeping SpO2 below 90% or if dyspnea does not improve, non-invasive positive pressure ventilation (NIPPV) may be offered at the discretion of the assistant team. NIPPV will be performed with the patient in a supine position at 45 degrees. The mask will be facial (oronasal or full face) with an appropriate size for each patient and adapted in a way to minimize leakage. A hydrocolloid dressing can be placed over the nose in order to avoid ulcerations and increase comfort. The NIPPV will be performed with the help of a ventilator with inspiratory and expiratory circuits or with Bilevel devices with a single circuit and exhalation valve according to the availability of each center.
  Other Names: NIV; Low flow Oxygen; Non-invasive positive pressure ventilation; Noninvasive positive pressure ventilation; Oxygen supplementation
  Arms: Standard respiratory support

SUMMARY:
Randomized clinical trial in which the main objective is to compare High Flow Nasal Cannula (HFNC) versus the standard respiratory care in the alleviation of dyspnea perception in patients with do-not-intubate (DNI) order. This is a pragmatic study that will take place in 10 Brazilians ICU facilities which are already participating in the main study RENOVATE NCT03643939.

DETAILED DESCRIPTION:
Do-not-intubate (DNI) is usually established in cases where endotracheal intubation (ETI) is considered disproportionate to prognosis and/or incompatible with the expression of wishes and values of the patient. Regardless of the profile of this care plan offered to patients with DNI, the control of dyspnea is one of its central objectives. The approach to dyspnea includes pharmacological measures such as opioids and non-pharmacological measures, such as oxygen therapy and Non-Invasive Ventilation, and more recently, the high flow nasal catheter (HFNC). HFNC provides high flow of heated and humidified mixed gas through a nasal cannula. In addition to the ability to generate high flows and supplemental oxygen, HFNC may generate a low level of positive airway pressure, may decrease dead space ventilation and may contribute to better patient comfort, such as the possibility of oral feeding while undergoing treatment, performing oral hygiene and allowing conversation and interaction with family members. This pilot study aims to evaluate the efficacy of HFNC in reducing dyspnea and improving comfort in patients with Acute Respiratory Failure (ARF) and DNI order.

ELIGIBILITY:
Inclusion Criteria:

Participants must be 18 years of age or older, with ARF of any cause on admission or post-extubation with prior DNI directives or DNI order determined in the current hospitalization.

Patients must meet the following criteria below:

1. Dyspnea (defined on the Borg scale ≥4);
2. SpO2 <90% or paO2 <60 mmHg in room air;
3. Absence of delirium;
4. One of the following:

A. Signs of respiratory distress and use of accessory muscles; B. Respiratory rate greater than 25 incursions per min .

Exclusion Criteria:

1. Refusal of treatment;
2. Agitation or non-cooperation;
3. Presence of delirium at the time of randomization;
4. Anatomical abnormalities that may interfere with the adjustment of the non-invasive positive pressure ventilation mask
5. Glasgow <12;
6. Psychomotor agitation that prevents adequate medical / nursing assistance requiring sedation;
7. Contraindications to NIV: uncontrollable vomiting, hypersecretion of the airways, facial deformities, trauma or extensive facial burn;
8. Presence of pneumothorax or extensive pleural effusion;
9. Expected imminent death, defined as an estimated death of less than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Dypnea | 48 hours
  Variation in dyspnea according to the Borg scale in 48 hours.

SECONDARY OUTCOMES:
Comfort | 48 hours
  Comfort measured in a visual analogue scale from 0-100
Dose of Opioid | 48 hours
  Cumulative dose of opioid
Delirium | 48 hours
  Cumulative Delirium rate measured by CAM-ICU
Intensive Care Unit (ICU) stay | 28 days
  total days inside the ICU
Mortality | 28 days
  Mortality in 28 days
Usage of respiratory support devices | 48 hours
  Total time in use of devices in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, MD, Study Director — Hospital do Coracao; Lara P Kretzer, MD, Principal Investigator — HU UFSC; Leticia Kawano-Dourado, MD, Principal Investigator — Hospital do Coracao; Israel S Maia, MD, Principal Investigator — Hospital do Coracao; Fernando Zampieri, MD, Study Chair — Hospital do Coracao
Locations (1):
- Hospital Nereu Ramos, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
under construction
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP and Informed Consent will be available in april 2021
Access Criteria: Publication